CLINICAL TRIAL: NCT06846723
Title: The Effect of Stress Ball on Pain, Anxiety, Satisfaction and Treatment Continuity in Patıents With Extracorporeal Shock Wave Lithotripsy
Brief Title: Stress Ball Effects to Pain, Anxiety, Satisfaction and Treatment Continuity During ESWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Canan KANAT, PhD, Department of Surgical Diseases Nursing, Principal investigator, Research assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinUESWL
Record Dates: First submitted 2025-01-28; First posted 2025-02-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Urolithiasis; Extracorporeal Shock Wave Lithotripsy
Keywords: stress ball; urolithiasis; ESWL; pain; anxiety
MeSH Terms: conditions — Urolithiasis; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: According to the randomization table, the information showing the patients included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU) and when the researcher (CK) goes to the patient for application, after filling out the "Informed Voluntary Consent Form", he will open the envelope and learn which group is in which group. Due to the nature of the study, patients and the researcher (CK) will not be blinded, since stress ball will be applied only to the patients included in the study. However, the researcher (EC) collecting the data will be blinded as he/she does not know which group the patients are in. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stress ball group (Experimental): In addition to the routine treatment and care practices of the outpatient clinic, the patients included in the study group will be applied stress ball during ESWL.
  Interventions: Other: Stress ball
- Control group (No Intervention): The control group will be received routine treatment and care in the unit.

INTERVENTIONS:
Other: Stress ball — In addition to the routine treatment and care practices of the outpatient clinic, the patients included in the study group will be applied stress ball during ESWL. The researcher (CK) will explain and show the patients how to apply the stress ball 10 minutes before the procedure. The stress ball will be applied during the ESWL session and a round, medium-hard, high-quality silicone ball with an average diameter of 6 cm will be used. Patients will be asked to take the ball in the palm of their hand and squeeze and release the ball once after counting to three. Patients will be instructed to continue this practice until the end of the ESWL procedure and to pay attention to the stress ball during the procedure. The ball will be washed and cleaned after each use and wiped with disposable asepsis wipes before being given to the patient.
  Arms: Stress ball group

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL), a minimally invasive procedure, is used in the treatment of urolithiasis. The shock waves used in this procedure, which does not require any incision, cause pain in the superficial structures of the body such as skin, muscles and deep structures such as costae, nerves and kidney tissue. This pain may cause patients not to tolerate the treatment, delay in recovery, decrease in the effectiveness of the treatment and decrease in satisfaction. Patients may also experience anxiety about the procedure prior to treatment. Anxious patients experience more pain during ESWL. Pain and anxiety increase the activation of the sympathetic nervous system and neuroendocrine response, leading to physiologic changes such as increased blood pressure, heart rate and oxygen requirement of the body. This may negatively affect the vital signs of the patients. Therefore, it is essential to relieve pain and anxiety in patients undergoing ESWL and pharmacologic and nonpharmacologic methods are used for this purpose. Pharmacologic methods such as analgesics, opioids and sedative agents are used to reduce pain and anxiety in patients. Since these methods have side effects such as nausea, vomiting, gastric bleeding, respiratory depression, tachycardia, constipation, the use of non-pharmacological methods that can be applied by nurses is increasing. One of the non-pharmacologic methods is the stress ball, which uses the sense of touch to divert attention with cognitive focus. In this simple, reliable, cheap and easily accessible method, pain and anxiety are reduced by directing the mind to the attention-grabbing stimulus.

DETAILED DESCRIPTION:
Urolithiasis, which affects more than 12% of the world population and is one of the most common diseases of the urinary system, is diagnosed with pain, urinary tract infection, hydronephrosis, colicky pain, hematuria, nausea, vomiting, fever and chills, foul-smelling and cloudy urine as a result of stone obstruction of the ureter. Extracorporeal shock wave lithotripsy (ESWL), which is a highly minimally invasive procedure, is used in the treatment of urolithiasis in case of failure of medical treatments. This method is particularly effective for renal stones smaller than 2 cm and located in the upper ureter; however, it is also frequently preferred before surgical intervention due to its noninvasiveness and low morbidity.

In extracorporeal shock wave lithotripsy, high-energy shock waves are used to break the stone into small pieces that can rapidly pass through the ureters. The shock waves used in this procedure, which does not require any incision, cause pain in superficial structures of the body such as skin, muscle and deep structures such as costae, nerves and renal tissue. This pain may cause patients not to tolerate the treatment, delay in recovery, decrease in the effectiveness of the treatment and decrease in satisfaction. In addition, patients may experience anxiety about the procedure to be performed before treatment. Patients who experience anxiety experience more pain during ESWL.

Pain and anxiety increase the activation of the sympathetic nervous system and neuroendocrine response, leading to physiologic changes such as increased blood pressure, heart rate and oxygen requirement of the body. This may negatively affect the vital signs of patients. Therefore, it is essential to eliminate pain and anxiety in patients undergoing ESWL and pharmacologic and nonpharmacologic methods are used for this purpose. Pharmacologic methods such as analgesics, opioids and sedative agents are used to reduce pain and anxiety in patients. Since these methods have side effects such as nausea, vomiting, gastric bleeding, respiratory depression, tachycardia, and constipation, the use of non-pharmacologic methods that can be applied by nurses is increasing. Stress ball, which is one of the non-pharmacologic methods, provides diversion of attention with cognitive focusing by using the sense of touch. In this simple, reliable, inexpensive and easily accessible method, pain and anxiety are reduced by directing the mind to the attention-grabbing stimulus. In the literature, studies evaluating the effect of music on pain and anxiety in patients undergoing ESWL are common; however, only two studies evaluating the effect of stress ball were found. In these studies, the effects of two different non-pharmacologic methods, both stress ball and music, were examined; however, the effects on the satisfaction levels of the patients and their attendance to ESWL sessions were not examined. In the literature, it was reported that approximately 72-75% of patients underwent three or more ESWL sessions at 7-10 day intervals. However, inadequate management of patients' pain and anxiety may adversely affect their continuity of treatment and cause them to prefer surgical intervention instead of continuing ESWL sessions. Based on this information, in this study, it was aimed to examine the effect of stress ball on pain and anxiety in patients undergoing ESWL, as well as the effect of stress ball on patients' satisfaction levels and ESWL continuation status, unlike the literature. With the findings of the study, it is planned to contribute to the literature and to provide evidence for the importance of the use of non-pharmacologic methods.

ELIGIBILITY:
Inclusion Criteria:

* Those who agreed to participate in the study and whose verbal and written consent was obtained,
* 18 years of age or older,
* Can speak, read and write Turkish,
* Does not have any cognitive, affective and verbal problems that prevent them from communicating,
* Open to communication,
* First time ESWL,
* The first session of ESWL will be administered,
* Body mass index <30 kg\m2,
* Have not taken any analgesic before the procedure,
* Not taking anticoagulants before the procedure,
* Have not experienced renal colic pain immediately before the procedure,
* Not pregnant,
* Patients for whom ESWL is not contraindicated for any reason will be included in the study.

Exclusion Criteria:

* No verbal or written authorization can be obtained,
* Under 18 years of age,
* They cannot speak, write or read Turkish,
* Have any cognitive, affective and verbal problem that prevents them from communicating,
* The one who is closed to communication,
* Previously undergone ESWL,
* You will undergo a second or more sessions of ESWL,
* Body mass index >30 kg\m2,
* Who has taken analgesics before the procedure,
* Anticoagulants taken before the procedure,
* Experiencing renal colic pain just before the procedure,
* Pregnant,
* Patients in whom ESWL is contraindicated will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Pain level | Up to six weeks
  Visual Analog Scale (VAS) will be used to determine the pain intensity of patients during and after ESWL procedure. VAS was developed to convert some values that cannot be measured numerically into numerical form. The VAS, which is an easy-to-understand, quick-to-use scale that allows meaningful comparison of measurements over time, consists of a 10 cm long line with subjective descriptive statements at both ends of the scale. The patient will be asked to place a mark on this 10 cm line indicating the level of pain during and after the ESWL procedure (0=No pain, 10=Unbearable pain). The distance from the beginning of the scale to the mark will be measured with a ruler and the pain level of the individual will be determined numerically in cm. A low score obtained from the VAS will indicate that the pain intensity of the individual is low/low and a high score will indicate that the pain intensity is high.
Anxiety level | Up to six weeks
  The State-Trait Anxiety scale, for which a Turkish validity-reliability study was conducted, will be used to determine anxiety levels before and after the procedure in patients undergoing ESWL. This scale was developed by Spielberger et al. in 1970 and can be applied to people over the age of 14. The scale consists of the State-Trait Anxiety Scale, which determines how the individual feels at a certain moment and condition, and the Trait Anxiety Scale, which determines how the individual feels regardless of the situation and condition. In the present study, the DAQ, which is structured to measure what is felt at that moment, will be used.

SECONDARY OUTCOMES:
Satisfaction level | Up to six weeks
  After the ESWL procedure, the satisfaction level of the patients with the ESWL procedure and their attendance to the next sessions will be recorded. Visual Analog Scale (VAS) was developed to convert some values that cannot be measured numerically into numerical form. VAS, which is a safe, easily applicable measurement tool generally accepted in the world literature, consists of a 10 cm long line with subjective descriptive statements at both ends of the scale. The patient will be asked to place a mark on this 10 cm line indicating the level of satisfaction with the ESWL procedure (0=Not at all satisfied, 10=Very satisfied).
Continuity of treatment | Up to six weeks
  The attendance of the patients to the next sessions will be checked from the follow-up list of patients undergoing ESWL in the outpatient clinic where the study was conducted and recorded on this form.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to avoid duplication, it is not intended to be shared until the research is completed.

REFERENCES:
- [Result] Browne C, Redmond E, Kelly T, Rogers E, O'Malley P, Nusrat N, Jaffry S, Durkan G, Walsh K, Dowling C, D'Arcy FT. Strategies to maximise patient comfort during extracorporeal shockwave lithotripsy - A randomised controlled trial. Surgeon. 2021 Aug;19(4):207-211. doi: 10.1016/j.surge.2020.07.002. Epub 2020 Aug 6. PMID 32771299
- [Result] 13. Torki, M., Heidari, H., Norian, K., Rabieie, L., & Sedehi, M. (2022). The effect of the distraction of thought by music on pain relief in patients undergoing extracorporeal shock wave lithotripsy: A randomized controlled trial. Journal of Shahrekord University of Medical Sciences, 24(2), 100-103.
- [Result] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283
- [Result] Ugras GA, Kanat C, Yaman Z, Yilmaz M, Turkmenoglu MO. The Effects of Virtual Reality on Preoperative Anxiety in Patients Undergoing Colorectal and Abdominal Wall Surgery: A Randomized Controlled Trial. J Perianesth Nurs. 2023 Apr;38(2):277-283. doi: 10.1016/j.jopan.2022.07.005. Epub 2022 Oct 29. PMID 36319521
- [Result] Duzel B, Cam Yanik T, Kanat C, Altun Ugras G. The effect of acupressure on pain level and hemodynamic parameters after coronary angiography: a randomized controlled study. Front Cardiovasc Med. 2023 Jul 14;10:1173363. doi: 10.3389/fcvm.2023.1173363. eCollection 2023. PMID 37522084
- [Result] Lei M, Li G, Tang Y, Yuan J, Yang T, Gao Z. Efficacy of music therapy for pain control of extracorporeal shock wave lithotripsy: A meta-analysis of randomized controlled studies. Medicine (Baltimore). 2024 May 31;103(22):e38182. doi: 10.1097/MD.0000000000038182. PMID 39259054
- [Result] Sokouti M, Sokouti M, Sokouti B. A systematic review and meta-analysis on the outcomes of extracorporeal shock wave compared to ureteroscopic lithotripsy for the treatment of ureteral stones. J Taibah Univ Med Sci. 2023 Jun 14;18(6):1459-1471. doi: 10.1016/j.jtumed.2023.06.001. eCollection 2023 Dec. PMID 37441243
- [Result] Gezginci E, Iyigun E, Yalcin S, Bedir S, Ozgok IY. Comparison of Two Different Distraction Methods Affecting the Level of Pain and Anxiety during Extracorporeal Shock Wave Lithotripsy: A Randomized Controlled Trial. Pain Manag Nurs. 2018 Jun;19(3):295-302. doi: 10.1016/j.pmn.2017.09.005. Epub 2017 Dec 14. PMID 29248604
- [Result] Chen HT, Hung KC, Hsu YC, Kuo JR, Chang YJ, Chen IW, Sun CK. Efficacy of acupuncture for pain relief in patients receiving extracorporeal shock wave lithotripsy: a meta-analysis of randomized controlled studies. Front Med (Lausanne). 2023 Jun 2;10:1114485. doi: 10.3389/fmed.2023.1114485. eCollection 2023. PMID 37332744